CLINICAL TRIAL: NCT01791725
Title: A 4-Week Randomized, Double-Blind, Placebo-Controlled, Phase 2a Safety and PK Study of Oral ELND005 in Young Adults With Down Syndrome Without Dementia
Brief Title: A 4-Week Safety Study of Oral ELND005 in Young Adults With Down Syndrome Without Dementia
Acronym: DS201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ELND005-DS201
Record Dates: First submitted 2013-02-06; First posted 2013-02-15 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — scyllitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ELND005 BID (Experimental): ELND005 250 mg BID
  Interventions: Drug: ELND005
- ELND005 QD (Experimental): ELND005 250 mg QD
  Interventions: Drug: ELND005
- Placebo (Placebo Comparator): Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ELND005
  Arms: ELND005 BID; ELND005 QD
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled, parallel-group, three-arm, multicenter study of the safety and PK of ELND005 administered orally for 4 weeks. This study will enroll Down Syndrome patients 18 to 45 years of age (inclusive) without dementia.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 45 years of age
* Has an IQ of > 40 (K-BIT)
* Able and willing to have a brain MRI

Exclusion Criteria:

* Symptoms of dementia or worsening cognition over the past year.
* Has a history of hepatitis B, hepatitis C, or HIV

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, San Diego, La Jolla, California
  - University of California, Irvine, Orange, California
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Rafii MS, Skotko BG, McDonough ME, Pulsifer M, Evans C, Doran E, Muranevici G, Kesslak P, Abushakra S, Lott IT; ELND005-DS Study Group. A Randomized, Double-Blind, Placebo-Controlled, Phase II Study of Oral ELND005 (scyllo-Inositol) in Young Adults with Down Syndrome without Dementia. J Alzheimers Dis. 2017;58(2):401-411. doi: 10.3233/JAD-160965. PMID 28453471

RESULTS

PARTICIPANT FLOW:
Groups:
- ELND005 BID: ELND005 250 mg BID
  ELND005
- ELND005 QD: ELND005 250 mg QD
  ELND005
- Placebo: Placebo BID
  Placebo
Period: Overall Study
Arm/Group | ELND005 BID | ELND005 QD | Placebo
Started | 12 | 5 | 6
Completed | 12 | 4 | 6
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ELND005 BID | ELND005 QD | Placebo | Total
Number analyzed (Participants) | 12 | 5 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (7.43) | 27.8 (4.03) | 30.0 (5.93) | 27.6 (6.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 9
  Male | 9 | 2 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 11 | 5 | 5 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 10 | 4 | 6 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 5 | 6 | 23
IQ Score [Mean (Standard Deviation); unit: units on a scale] — IQ was measured by the Kaufman Brief Intelligence Test (KBIT)
  units on a scale | 50.6 (13.81) | 63.3 (19.62) | 55.8 (6.65) | 54.3 (13.75)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (TEAEs)
Description: For all AE summaries, if a patient had more than one AE within a preferred term, the patient was counted only once, at the maximum severity and with the closest relationship to study drug. If a patient had more than one AE within a SOC, the subject was similarly counted only once when reporting results for that SOC.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | ELND005 BID | ELND005 QD | Placebo
Number analyzed (Participants) | 12 | 5 | 6
participants | 5 | 2 | 0

2. Other Pre Specified Outcome: Changes From Baseline in Abnormal Neurological Examination Results
Description: Subjects with Abnormal Neurological Examination Results
Time Frame: Baseline and 4 weeks
Measure: Number; unit: participants
Arm/Group | ELND005 BID | ELND005 QD | Placebo
Number analyzed (Participants) | 12 | 4 | 6
participants
  Baseline | 4 | 1 | 3
  Week 4 | 4 | 1 | 3

3. Other Pre Specified Outcome: Pharmacokinetic Assessment
Description: Mean Plasma ELND005 Concentrations- Cmax
Time Frame: Baseline and 4 Weeks
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | ELND005 BID | ELND005 QD | Placebo
Number analyzed (Participants) | 12 | 4 | 6
μg/mL
  Mean Cmax, First Dose, Day 0 | 1.68 (0.90) | 2.61 (0.62) | 0 (0)
  Mean Cmax, Last Dose, Day 28 | 6.33 (1.95) | 4.48 (1.13) | 0 (0)

4. Other Pre Specified Outcome: Cognitive Outcome (RADD Total Score)
Description: Rapid Assessment for Development Disabilities (RADD) The RADD test was developed from the low-difficulty items from published intelligence tests (Walsh et al 2007). It was specifically developed for evaluation of individuals with intellectual disabilities and developmental disabilities. It is a validated and reliable cognitive screening instrument that can be rapidly administered. The RADD is composed of 76 items. Each item is scored as 0 (incorrect) or 1 (correct).The test assesses a wide range of functional abilities including receptive and expressive language, orientation, registration, recall, attention, self identification, motor skills, imitation, abstract reasoning, number skills, comprehension and short-term memory to give a total score. Scores are from 0 to 76. A higher total score is correlated with a higher Cognitive Impairment level.
Time Frame: Baseline and 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ELND005 BID | ELND005 QD | Placebo
Number analyzed (Participants) | 12 | 4 | 6
units on a scale
  Day 0 | 58.7 (10.2) | 58.0 (15.6) | 62.2 (9.8)
  Week 4 | 59.1 (11.5) | 64.3 (13.5) | 62.8 (10.3)

5. Other Pre Specified Outcome: Improvement in NPI Total Scores in Subjects With NPI Score ≥1 at Baseline Baseline
Description: The Neuropsychiatric Inventory(NPI) (Cummings et al 1994) is a behavioral measure that assesses psychopathology in dementia patients. The NPI was administered at the Baseline Visit (Day 1) and at Day 28 (EOS) or ET. A decrease in score shows an improvement in symptoms.
Time Frame: Baseline and 4 weeks
Population: Subjects with NPI Score ≥1 at baseline
Measure: Number; unit: participants
Arm/Group | ELND005 BID | ELND005 QD | Placebo
Number analyzed (Participants) | 8 | 4 | 3
participants | 7 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for each patient, starting from the time the consent form was signed until completion of the study.
Arm/Group | ELND005 BID | ELND005 QD | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 5/12 | 2/5 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELND005 BID (N=12) | ELND005 QD (N=5) | Placebo (N=6)
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Catheter Site Pain (General disorders) | 0 | 1 | 0
Seasonal Allergy (Immune system disorders) | 1 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Resting Tremor (Nervous system disorders) | 1 | 0 | 0
Anger (Psychiatric disorders) | 0 | 1 | 0
Pseudofolliculitis barbae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Oral Disorder (Gastrointestinal disorders) | 1 | 0 | 0
Restless leg syndrome (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days